CLINICAL TRIAL: NCT02861612
Title: Nerve Transfers to Restore Hand Function in Spinal Cord Injury
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient patient recruitment
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Neurotrauma Foundation (Other); Canadian Society of Plastic Surgeons (Other); Washington University School of Medicine (Other); Rick Hansen Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 5313
Record Dates: First submitted 2016-07-13; First posted 2016-08-10 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Quadriplegia; Spinal Cord Diseases; Spinal Cord Injuries
Keywords: peripheral nerves; quadriplegia; nerve transfer; surgical procedures, operative; hand; upper extremity; quality of life
MeSH Terms: conditions — Quadriplegia; Spinal Cord Diseases; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nerve Transfer: This is an observational study that looks at function and quality of life in patients before and after nerve transfer surgery.
  Interventions: Procedure: Nerve Transfer Surgery

INTERVENTIONS:
Procedure: Nerve Transfer Surgery — Unilateral surgery will be performed under general non-paralytic anesthesia and no-tourniquet conditions to allow for responsive nerve simulation.

SUMMARY:
This study seeks to evaluate the efficacy of nerve transfers in restoring hand function in patients with cervical spinal injuries.

DETAILED DESCRIPTION:
Cervical spinal cord injury is a life-altering injury that results in profound loss of upper limb function. Hand function is essential to basic activities of daily living and consequently has a significant impact on patients' quality of life. Tendon transfers and/or tenodesis have traditionally been used to restore hand function in spinal cord injuries - however, in recent years there is growing interest in the role of nerve transfers as a means of accomplishing this goal. Although preliminary results indicate nerve transfers may be well-suited for patients with spinal cord injury, their long term efficacy has not been demonstrated.

This study seeks to evaluate the efficacy of nerve transfers in restoring hand function in patients with cervical spinal injuries. Eligible patients will receive nerve transfer procedure(s) (e.g. brachialis to anterior interosseous nerve, supinator to posterior interosseous) and will be followed post-operatively to assess for changes in strength, functional independence, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a spinal cord injury AIS level C5 to C7. Those with motor complete injuries (AIS A or B) will be considered for surgical intervention if they are ≥ 5 months post injury. Motor incomplete patients (AIS C or D) will be considered if they are ≥ 1.5 years post injury.
* Patients will require ≥ MRC 4 strength of the muscle supplied by the donor nerve (e.g. brachialis, supinator).
* Finger flexor and extensor strength should be ≤ MRC 1 strength.
* Muscles supplied by the donor nerve, will need to have no or minimal of evidence of lower motor neuron injury as dictated by evidence of fibrillations, positive sharp waves, or moderate or severely decreased recruitment on needle electromyography.
* Those being evaluated for surgery outside nine-months post injury recipient muscles will be required to be free of lower motor neuron pathology.
* Ability to comply and participate in rigorous post-surgical therapy regimen.

Exclusion Criteria:

* Comorbidities precluding safe surgery including autonomic/hemodynamic instability, pulmonary instability, active infection, chronic pressure sores or untreated urinary tract infections as determined by physician.
* Simultaneous tendon transfer or tenodesis surgery (which would preclude separation of the effect of nerve transfer alone).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Any patients with cervical spinal cord injury and upper extremity dysfunction who are medically stable, residents of Canada, willing and able to be assessed at the The Ottawa Hospital are potential participants.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2019-03-18 (Estimated); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Upper extremity function - Myometric measures of strength (donor and recipient muscle groups) | Change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  Valid and reliable quantitative muscle strength measurement
Upper extremity function - Manual muscle testing (MRC) | Change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  Quantitative assessment of motor function (MRC)
Upper extremity function - Graded Redefined Assessment of Strength, Sensibility and Prehension test (GRASSP) | Change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  Valid, reliable and responsive measure of sensorimotor upper limb impairment specifically designed for patients with cervical SCI
Upper extremity function - Range of motion | Change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  Quantitative assessment of range of motion (degrees)

SECONDARY OUTCOMES:
Health related quality of life - The Short Form (SF)-36 | Change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  Valid and responsive measure of quality of life in surgical patients
Health related quality of life - Spinal Cord Independence Measure (SCIM I) | Change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  Disability scale developed to specifically address the ability of SCI patients to perform basic activities of daily living independently
Health related quality of life - Canadian Occupational Performance Measure (COPM) | Change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  Evidence-based outcome measure designed to capture a patient's self-perception of performance in everyday living
Health related quality of life - Semi-structured interviews | Collected at 12 and 24 months post-surgery.
  Semi-structured interviews to gain information about satisfaction, acceptability, and the subjective experience of the surgical intervention, therapy, and functional outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty U Boyd, MD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Washington University School of Medicine, St Louis, Missouri, United States
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Nerve Transfers to Restore Upper Extremity Function in Cervical Spinal Cord Injury: Update and Preliminary Outcomes. Plast Reconstr Surg. 2015 Oct;136(4):780-792. doi: 10.1097/PRS.0000000000001641. PMID 26397252
- [Background] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Use of peripheral nerve transfers in tetraplegia: evaluation of feasibility and morbidity. Hand (N Y). 2015 Mar;10(1):60-7. doi: 10.1007/s11552-014-9677-z. PMID 25767422